CLINICAL TRIAL: NCT00005070
Title: A Phase II Trial of 6-Hydroxymethylacylfulvene (HMAF; MGI-114) in Patients With Advanced Cervical Carcinoma
Brief Title: Irofulven in Treating Patients With Stage IVB or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-072; CDR0000067675 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0096
Record Dates: First submitted 2000-04-06; First posted 2004-08-09 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irofulven in treating patients who have stage IVB or recurrent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of 6-hydroxymethylacylfulvene in patients with stage IVB or recurrent cervical carcinoma. II. Determine the safety of this drug in this patient population.

OUTLINE: Patients receive 6-hydroxymethylacylfulvene IV over 5 minutes daily for 5 consecutive days. Treatment continues every 28 days in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 6-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary metastatic (stage IVB) or recurrent cervical carcinoma not amenable to curative therapy Squamous Adenocarcinoma Adenosquamous Bidimensionally measurable disease No active brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal ALT/AST no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN (1.95 mg/dL at MSKCC) OR Creatinine clearance at least 50 mL/min Cardiovascular: No New York Heart Association class III or IV congestive heart failure No ECG evidence of acute ischemia No significant conduction abnormality (e.g., bifascicular block, 2nd or 3rd degree AV blocks) Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other malignancy within the past 5 years and deemed low risk for recurrence No other concurrent clinical circumstances that would compromise safety or integrity of trial

PRIOR CONCURRENT THERAPY: Prior multimodality therapy at diagnosis allowed (i.e., concurrent chemotherapy and radiotherapy, neoadjuvant chemotherapy followed by surgery and/or radiotherapy, adjuvant chemotherapy and/or radiotherapy following surgery, or adjuvant chemotherapy following radiotherapy) Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic or recurrent disease Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 4 weeks since prior major surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Aghajanian, MD, Study Chair — Memorial Sloan Kettering Cancer Center